CLINICAL TRIAL: NCT06871293
Title: Impact of Functional and Cognitive Rehabilitation, in Adults with Chronic Noncommunicable Diseases and Long Covid-19 , on Their Functional and Cognitive Capacity, Quality of Life, and the Evolution of Their Baseline Condition, in Bogotá D.C.
Brief Title: Evaluating the Impact of a Functional and Cognitive Strategy in Patients with Long Covid-19
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Cardioinfantil Instituto de Cardiología (Other)
Collaborators: Hospital Militar Central, Colombia (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024PROEPI0164; ATENEA-366-2022 (Other Grant/Funding Number: Agencia Distrital para la Educación Superior, la Ciencia y la Tecnología-ATENEA)
Record Dates: First submitted 2025-03-05; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Long COVID-19 Syndrome; COVID 19; Noncommunicable Disease; Hypertension; Diabetes Mellitus; Long COVID
Keywords: Covid 19; Sars CoV 2; Post-acute Covid-19 syndrome; Long Covid; Hypertension; Diabetes Mellitus; Noncommunicable disease; Rehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome; COVID-19; Noncommunicable Diseases; Hypertension; Diabetes Mellitus | interventions — Functional Status

STUDY DESIGN:
Intervention Model Description: Parallel-group, randomized controlled trial (RCT) with active control.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Functional and Cognitive Rehabilitation (Active Comparator): Participants assigned to the functional and cognitive rehabilitation strategy will attend one weekly session for 8 weeks at study sites. Each session includes one hour of functional rehabilitation (warm-up, aerobic exercise, muscle strengthening, and cool-down) supervised by healthcare professionals who monitor effort levels and heart rate. Additionally, participants will receive 30 minutes of cognitive rehabilitation, focusing on memory, attention, and executive functions, guided by occupational therapists or speech therapists. This intervention aims to enhance physical and cognitive function in patients with chronic diseases and Long Covid-19.
  Interventions: Other: Evidence-Based Informational Support
- Evidence-Based Informational Support (Active Comparator): Participants assigned to the evidence-based informational support arm will receive weekly educational messages for 8 weeks via email or text messages. These messages are derived from a thorough review of high-quality scientific studies and cover key topics related to Covid-19 prevention, treatment, follow-up, and prognosis. A total of 24 informational pieces will be delivered, ensuring patients receive clear, research-based guidance to support their health management. This intervention aims to improve patient awareness and self-care strategies for Long Covid-19 and chronic conditions.
  Interventions: Other: Functional and cognitive rehabilitation strategy

INTERVENTIONS:
Other: Functional and cognitive rehabilitation strategy — The functional and cognitive rehabilitation strategy is a structured, supervised program, designed to improve physical and cognitive function in patients with Long Covid-19 and chronic diseases. Participants will attend weekly in-person sessions for 8 weeks at study sites.
  Each session includes:
  * Functional Rehabilitation (60 min): Warm-up, aerobic exercise (elliptical/treadmill), muscle strengthening, and cool-down, all supervised by trained healthcare professionals who monitor effort levels and heart rate.
  * Cognitive Rehabilitation (30 min): Memory, attention, and executive function exercises, guided by occupational therapists or speech therapists.
  Arms: Evidence-Based Informational Support
Other: Evidence-Based Informational Support — The evidence-based informational support intervention provides structured, research-based health information to patients with Long Covid-19 and chronic diseases. Participants receive weekly digital messages for 8 weeks via email or text, covering key topics such as Covid-19 prevention, treatment, follow-up, and prognosis.
  Content is derived from high-quality scientific studies and clinical guidelines.
  A total of 24 informational pieces are delivered, ensuring comprehensive coverage of essential health recommendations.
  This intervention is remote, accessible, and designed to enhance patient knowledge and self-management, distinguishing it from traditional in-person education programs.
  Arms: Functional and Cognitive Rehabilitation

SUMMARY:
This study aims to evaluate the impact of a functional and cognitive rehabilitation strategy compared to evidence-based informational messages, on functional capacity, cognitive abilities, quality of life, and disease progression in adults with chronic non-communicable diseases (NCDs) and Long Covid-19.

Researchers will compare a structured rehabilitation program to informational support through evidence-based messages to determine if rehabilitation leads to better functional and cognitive outcomes in patients with Long Covid-19.

Participants will be randomly assigned to one of two groups:

1. Functional and cognitive rehabilitation: Attending weekly in-person sessions for 8 weeks, including supervised physical and cognitive exercises.
2. Informational support: Receiving weekly evidence-based educational messages for 8 weeks.

Participants will undergo assessments at baseline, post-intervention, and six months later, including a six-minute walk test, handgrip strength measurement, and questionnaires on disability, anxiety, depression, fatigue, dyspnea, cognitive function, and quality of life.

DETAILED DESCRIPTION:
Study Objective

The primary goal of this study is to evaluate the impact of a functional and cognitive rehabilitation strategy compared to evidence-based informational messages, on functional capacity, cognitive abilities, quality of life, and disease progression in adults with chronic non-communicable diseases (NCDs) and Long Covid-19.

Specific Objectives

* Determine the prevalence of Long Covid-19 among participants from previous Covid-19 institutional registries, describing the primary clinical manifestations based on symptom recurrence and severity.
* Administer a functional and cognitive rehabilitation strategy in patients with NCDs and Long Covid-19, and compare it with evidence-based informational messages

Evaluate the impact of both interventions on key clinical outcomes, including:

* Six-minute walk test performance (functional capacity)
* Montreal Cognitive Assessment (MoCA) score (cognitive function)
* EQ-5D-5L (quality of life assessment)
* Incidence of events indicating worsening of underlying conditions

Methodology

The study has been conducted in two phases. The second phase is the one being registered on this platform:

1. Phase 1: Identification and Diagnosis of Long Covid-19

   * Study Design: Identification of eligible patients through institutional registries at Fundación Cardioinfantil - Instituto de Cardiología (FCI-IC) and Hospital Militar Central (HOMIL).
   * Eligible Population: Adults (≥18 years) with a history of hypertension or type 2 diabetes mellitus who had a suspected acute SARS-CoV-2 infection between March 2020 and December 2021.
   * Sample Size and Recruitment: Approximately 2,240 individuals were contacted, with an expected 30% prevalence of long COVID, yielding at least 672 eligible participants for the clinical trial.

   Screening Procedures:
   * Telephone contact using a pre-established script adapted from one of the registries.
   * Administration of a structured questionnaire on persistent symptoms, functional limitations, and prior health conditions.

   Criteria for Long Covid-19 diagnosis:
   * Presence of at least two persistent, intermittent, or recurrent symptoms for at least four weeks.
   * At least one symptom significantly impacting daily activities.
   * Symptoms unexplained by pre-existing health conditions.

   Data Management: Information has been recorded in the REDCap platform, ensuring secure data collection and monitoring.
2. Phase 2: Randomized Clinical Trial

   * Study Design: A parallel-group, randomized controlled trial (RCT) with active control.
   * Eligible Participants: Those diagnosed with Long Covid-19 in Phase 1.

Randomization (1:1):

* Experimental Group: Functional and cognitive rehabilitation strategy.
* Control Group: Informational support with evidence-based messages.

Inclusion Criteria:

* Confirmed Covid-19 diagnosis.
* History of hypertension or diabetes before the SARS-CoV-2 infection.
* Persistent symptoms affecting daily life.
* Ability to participate in in-person rehabilitation or receive informational support.

Exclusion Criteria:

* Age >80 years.
* Advanced chronic conditions (e.g., severe heart failure, advanced kidney disease).
* Hospitalizations in the year prior to study enrollment.
* Cognitive or physical impairments preventing participation.
* Interventions

Functional and Cognitive Rehabilitation:

Duration: 8 weeks, with one session per week at the study site.

1. Functional Rehabilitation (Supervised by trained health professionals)

   * Warm-up (8 min)
   * Aerobic exercise (20 min on treadmill/elliptical)
   * Muscle toning (8 min)
   * Cool-down (8 min)
2. Cognitive Rehabilitation (Guided by occupational therapy professionals) - 30-minute sessions focusing on memory, attention, and executive functions.

Informational Support with evidence-based messages (Active Control):

Weekly delivery of evidence-based health information via email, SMS, or WhatsApp. Topics include COVID-19 prevention, treatment, and prognosis.

Three informational messages per week for 8 weeks.

Outcome Measures

1. Primary Outcomes:

   * Six-minute walk test.
   * MoCA cognitive assessment.
   * EQ-5D-5L quality of life questionnaire.
   * Incidence of clinical events related to NCD deterioration.
2. Secondary Outcomes:

   * Fatigue severity (Fatigue Severity Scale).
   * Anxiety and depression (Hospital Anxiety and Depression Scale).
   * Disability assessment (WHO Disability Assessment Schedule 2.0).
   * Dyspnea severity (MRC Dyspnea Scale).

Additionally, complementary measurements will be taken at the initial visit, post-intervention, and six months after completion to assess:

* WHO Disability Assessment Questionnaire.
* Hospital Anxiety and Depression Scale.
* Fatigue Severity Scale.
* MRC Dyspnea Scale.
* Study Timeline and Follow-up Baseline assessment (before intervention).
* Post-intervention evaluation (within 4 weeks of completion).
* Six-month follow-up assessment.
* Evaluations conducted by trained, blinded assessors to ensure objectivity.

Ethical Considerations

* Confidentiality: Participant data will be managed per ethical guidelines and stored securely.
* Voluntary Participation: Participants may withdraw without affecting their standard medical care.
* Safety Measures: Rehabilitation sessions will be supervised to mitigate risks such as fatigue or dizziness.
* Insurance Coverage: A study-specific insurance policy will provide coverage for any adverse events related to the interventions.

This study will contribute to understanding Long Covid-19 management in patients with chronic conditions, providing evidence for the development of effective rehabilitation strategies to improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Covid-19 confirmed.
* History of arterial hypertension or diabetes mellitus before entering the institutional registries of the FCI-IC or HOMIL, institutional registries of the FCI-IC or HOMIL or before having the diagnosis of SARSCoV-2 infection.
* Persistence of two or more concurrent symptoms, related to Covid-19 prologue, for at least 4 weeks (persistent, intermittent, or intermittent).
* At least one of these symptoms must have an impact on activities of daily living. They can be physical (fatigue, dyspnea, myalgias, arthralgias) or neuropsychiatric (cognitive, sleep and emotional alterations).
* Symptoms unexplained by underlying disease or other condition concomitant with SARS-CoV-2 infection. SARS-CoV-2 infection (determined by prior medical history review and participant interview).

participant interview).

- Ability to read and attend functional and cognitive rehabilitation sessions or to receive the with evidence-based informational messages.

Exclusion Criteria:

* Age >80 years.
* Severely advanced baseline comorbidities prior to SARS-CoV-2 infection.
* Presence of chronic respiratory disease (partial or permanent supplemental oxygen use), cardiac failure (LVEF<40%) or advanced renal disease (GFR<30%).

heart failure (LVEF<40%) or advanced renal disease (GFR<30).

* Two hospitalizations in the year prior to admission to the institutional registries of the FCI-IC and the HOMIL for the patient's underlying disease.
* Dependence on a caregiver.
* Orthopedic or cardiopulmonary problems that contraindicate the performance of aerobic exercise.
* Neuropsychiatric or cognitive limitations that limit understanding or following commands and performing attention exercises.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Composite Change in Functional Capacity, Cognitive Function, Health-Related Quality of Life, and Strength | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  The primary outcome is a composite measure evaluating the aggregated change across four key functional and cognitive scales:
  * Functional Capacity with six-minute walk test.
  * Cognitive Function with Montreal Cognitive Assessment, MoCA. The minimum score is 0 points, which would indicate very severe cognitive impairment, since the maximum total score is 30 points. Normally, a score of 26 or higher is considered within the normal range, although the range may vary depending on factors such as the patient's age and educational level. A score below 26 could suggest possible cognitive impairment, and the lower the score, the more indicative it may be of severe cognitive problems.
  * Health-Related Quality of Life with EuroQol 5 Dimensions 5 Levels, EQ-5D-5L. Maximum value: 1 This value corresponds to the best possible health state. Minimum value: -0.594 This value corresponds to the worst possible.
  * Handgrip Strength with hydraulic dynamometer.

SECONDARY OUTCOMES:
Change in Functional Capacity | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  Distance covered in six minutes will be measured and compared to baseline values. Additional tests include the four-step climb power test and the 30-second sit-to-stand test, evaluating lower body strength and endurance.
  Greater distance indicates better functional capacity. Lower values may indicate physical dysfunction or a chronic illness.
Change in Cognitive Function | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  Montreal Cognitive Assessment scores will be used to assess changes in memory, visuospatial abilities, executive function, attention, language, and orientation.
  The minimum score is 0 points, which would indicate very severe cognitive impairment, since the maximum total score is 30 points. Normally, a score of 26 or higher is considered within the normal range, although the range may vary depending on factors such as the patient's age and educational level. A score below 26 could suggest possible cognitive impairment, and the lower the score, the more indicative it may be of severe cognitive problems.
Change in Health-Related Quality of Life | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  Changes in mobility, self-care, usual activities, pain/discomfort, and anxiety/depression will be evaluated using EuroQol 5 Dimensions 5 Levels.
  Maximum value: 1 This value corresponds to the best possible health state. Minimum value: -0.594 This value corresponds to the worst possible.
Change in Health-Related Quality of Life, Visual Analogue Scale | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  In addition to the score based on the 5 dimensions, the VAS scale from 0 to 100, where: 0 represents the worst imaginable health and 100 represents perfect health.
Change in Handgrip Strength, Hydraulic Dynamometer | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  Bilateral handgrip strength will be measured according to the American Society of Hand Therapists guidelines. Changes in dominant and non-dominant hand strength will be assessed.
Incidence of Chronic Disease Decompensation Events | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  Participants will report new medical visits, hospital admissions, medication adjustments, or cardiovascular events related to their underlying chronic condition.
Additional Functional and Clinical Assessments | Baseline (Day 1), 4 weeks post-intervention, and 6-month follow-up.
  Complementary assessments will be conducted at baseline, post-intervention, and six-month follow-up, including:
  * WHO Disability Assessment Schedule 0-24: No significant disability 25-49: Mild to moderate disability 50-74: Moderate to severe disability 75-100: Severe or extreme disability
  * Hospital Anxiety and Depression Scale 0-7 points: Normal, no signs of anxiety or depression. 8-10 points: Possible signs of anxiety or depression, follow-up is needed. 11-21 points: Indicative of clinically significant symptoms of anxiety or depression, suggesting a more detailed evaluation is needed.
  * Fatigue Severity Scale
    1 - 3: Low fatigue 4 - 5: Moderate fatigue 6 - 7: Severe fatigue
  * Medical Research Council Dyspnea Scale Level 1: No difficulty breathing during normal activities. Level 2: Dyspnea with moderate physical activities. Level 3: Dyspnea with everyday physical activities. Level 4: Dyspnea with minimal exertion. Level 5: Dyspnea at rest, indicating sever

CONTACTS AND LOCATIONS:
Locations (1):
- Fundación Cardioinfantil-Instituto de cardiología, Bogotá DC, Bogotá DC, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
Data from the study would be provided by request to the principal investigator